CLINICAL TRIAL: NCT01292772
Title: The Effects of Radiation Therapy on the Reconstructed Breast: An Evaluation Using MR Imaging
Brief Title: The Effects of Radiation in Reconstructed Breasts
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 12110
Record Dates: First submitted 2011-02-01; First posted 2011-02-10 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: breast cancer; bilateral mastectomy; immediate breast reconstruction; locally advanced unilateral breast cancer; bilateral mastectomy for prophylaxis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: contract-enhanced MRI — Patients will have contrast-enhanced MRI of the breasts.
Radiation: Unilateral Adjuvant Radiation Therapy — The study group will consist breasts receiving post-operative radiation, and the control group will consist of the patient's breasts on the non-radiated side. In this way, patients will act as their own control.

SUMMARY:
The primary objective of this study is to use LR imaging to evaluate the effects of adjuvant radiation therapy on reconstructed breasts.

DETAILED DESCRIPTION:
Immediate breast reconstruction following mastectomy has become an increasingly popular and accepted treatment option among breast cancer patients. This change in practice has resulted in a significant number of patients who undergo radiation therapy after breast reconstruction. Following irradiation, the reconstructed breast often experiences fibrotic contracture, volume loss, altered pigmentation, or some combination thereof, producing an asymmetric and aesthetically compromised result. The effects of radiation on reconstructed breasts as well as the implications that such changes have for timing of reconstructive surgery, post-operative management and surveillance imaging are topics of growing importance in plastic surgery, radiology and surgical oncology.

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18 and 90 years of age.
* Patients with a diagnosis of unilateral breast cancer who elect to undergo bilateral mastectomy with immediate free flap reconstruction.
* Patients must also have a locally advanced tumor that requires adjuvant radiation therapy following reconstruction.

Exclusion Criteria:

* Women who do not undergo immediate, bilateral breast reconstruction using a free flap.
* Women who do not require unilateral, adjuvant radiation therapy
* Women who are pregnant
* Women who have altered renal function, defined as a personal history of diabetic, hypertensive or autoimmune nephropathy and/or on routine preoperative testing are found to have a serum creatinine greater than or equal to 1.3

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will consist of patients with a diagnosis of unilateral breast cancer who elect to undero bilateral mastectomy with immediate free flap reconstruction. Patients will be treated by members of the Division of Plastic and Reconstructive Surgery and will receive postoperative radiation therapy to the affected breast.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Reconstructed Breast Volume | up to 1 year after radiation
  This will be compared at 2 points: before radiation and 1 year after radiation is completed between the 2 breasts.
Vascular Fibrosis | up to 1 year after radiation
  This will be compared at 2 points: before radiation and 1 year after radiation is completed between the 2 breasts.
Dermal Thickness | up to 1 year after radiation
  This will be compared at 2 pionts: before radiation and 1 year after radiation is completed between the 2 breasts

SECONDARY OUTCOMES:
Presence of Fat Necrosis in the Breast | up to 1 year after radiation
  This will be assessed at 2 points: before radiation and 1 year after radiation is completed between the 2 breasts.
Evidence of Cancer Recurrence | up to 1 year after radiation
  This will assessed at 2 points: before radiation and 1 year after radiation is completed between the 2 breasts.
Symmetry | up to 1 year after radiation
  This will be assessed at 2 points; before radiation and 1 year after radiation is completed between the 2 breasts.
Hyperpigmentation | up to 1 year after radiation
  This will be assessed at 2 points: before radiation and 1 year after radiation is completed between the 2 breasts.
Contracture | up to 1 year after radiation
  This will be assessed at 2 points:before radiation and 1 year after radiation is completed between the 2 breasts.
Aesthetic Result | up to 1 year after radiation
  This will be assessed at 2 points: before radiation and 1 year after radiation is completed between the 2 breasts.

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States